CLINICAL TRIAL: NCT02486341
Title: Daily Glycaemic Variability in Frail or Disabled Older Patients With Diabetes Over 75 Treated With Basal Insulin
Acronym: VARQUOGLY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CHUBX 2014/08
Record Dates: First submitted 2015-06-09; First posted 2015-07-01 (Estimated); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Diabetes
Keywords: continuous glucose monitoring system; basal insulin; diabetes mellitus; elderly
MeSH Terms: conditions — Diabetes Mellitus | interventions — Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Human Neutral Protamine Hagedorn (NPH) (Experimental): The inclusion will be stratified into 2 groups according to the type of basal insulin being at baseline (ratio 1: 1): NPH human insulin / Long-acting basal insulin analogues. The type of insulin will not be changed by this protocol.
  Interventions: Drug: Insulin
- Long-acting basal insulin analogues (Experimental)
  Interventions: Drug: Insulin

INTERVENTIONS:
Drug: Insulin — Continuous glucose monitoring system over 120-hour period.

SUMMARY:
Basal insulin is widely used in older patients with diabetes. Human insulin Neutral Protamine Hagedorn (NPH) has been proposed as basal insulin in older (75 years or older) frail and dependent patients due to its shorter action. However, no study has analysed the glycaemic profile in elderly subjects according to the basal insulin used, particularly in frail or disabled patients.

The aim of this study is to measure intra-day glycaemic variability according basal insulin (human NPH or long acting analogues) in older (75 and older) frail or disabled patients with diabetes using continuous glucose monitoring system.

DETAILED DESCRIPTION:
Increased prevalence of diabetes mellitus is in large part related to ageing: in France in 2009, 26% of patients with diabetes were 75 older or over. Moreover, diabetes prevalence is particularly high among institutionalized subjects with more than half of them treated with insulin.

Diabetes is source of activities limitations and participation restriction from the early stages of the disease and is responsible for 10% of direct health costs, with higher costs for older patients or insulin treated patients.

Older patients with diabetes may be robust (fully independent), frail or disabled. Studies with patients of 75 years or older included mainly robust subjects. Nevertheless older patients with diabetes are more frequently frail and a large proportion have a different metabolic profile than younger ones: they are leaner and present more often with beta-cellular insufficiency. Frail or dependent patients may also have different nutritional status than robust ones. Thus, this is difficult to extrapolate what is known about glycaemic profile in robust and young older (65-74 years old) insulin-treated patients to frail and dependent older ones (>74 years).

Continuous blood glucose monitoring systems give the opportunity to measure around the day the blood glucose variations in real-life and particularly nocturnal hypoglycaemia for these patients treated with various types of basal insulins.

ELIGIBILITY:
Inclusion Criteria:

* Age> or equal to 75 years,
* Diabetes mellitus diagnosed or Glycated hemoglobin (HbA1c) > 7% or 2 fasting blood glucose > to 1.26g/l,
* Treated with basal insulin associated or not with metformin (one or two injections per day, in the morning and/or evening before meals)
* Subject affiliated or beneficiary of a social security system,
* Free consent, informed and signed by the participant or by the surrogate of the patient and the investigator,
* Patient in the 4th or higher categories of frailty according to Rockwood .

Exclusion Criteria:

* Refusal of wearing a continuous glucose monitoring system,
* Total autonomy (mobility according to Rosow and Breslau scale, instrumental activities of daily living according to Lawton scale, activities of daily living according to Barthel score),
* Treatment with insulinosecretors Dipeptidyl peptidase-4 inhibitor, Glucagon-like peptide-1 analogues, sulfonylurea) or rapid insulin (human or rapid analogue),
* Daily dose of basal insulin with change of 20% or more in the last 7 days,
* Current treatment with corticosteroids,
* Acute pathology in the last 7 days :
* Infection treated with antibiotic
* New stroke in the last 7 days
* Cardio-respiratory decompensation: change in daily dose of diuretics or oxygenotherapy during the last 7 days,
* Clinically unstable patients according judgement of investigator,
* Behavioural disturbances like Agitation/Aggressivity according the Neuropsychiatric Inventory (NPI),
* All people who are under legal protection,
* All people who will be not able to finish the follow of the study,
* Currently participating in another clinical trial investigating.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-03-31 (Actual); Primary Completion 2019-01-28 (Actual); Study Completion 2019-01-28 (Actual)

PRIMARY OUTCOMES:
Intraday glycemic variability measured by the average of MAGE index (Mean amplitude of glycemic excursions) everyday of exploitable recording by the participant. | 5 days

SECONDARY OUTCOMES:
Intraday glycemic variability measured by the average standard deviation of blood glucose every day of exploitable recording by the participant | 5 days
Inter-day glucose variability assessed by Mean Differences of Daily per participant for every day of exploitable recording | 5 days
Average number of diurnal hypoglycaemia defined by blood glucose <0.60g / l from 7am to 22 pm for all exploitable recording days | 5 days
Average number of nocturnal hypoglycemia, defined by blood glucose < 0.60g / l between 22h and 7h for every day of exploitable recording | 5 days
Average time (minutes / day) per day pass in hypoglycemia (<0.60g / l) | 5 days
Nutritional status: a composite outcome measure consisting of multiple measures with Mini Nutritional Assessment, calf circumference, abdominal circumference, albumin | At inclusion
Functional Status: a composite outcome measure consisting of multiple measures with scale Rosow and Breslau, Lawton Instrumental Activities of Daily Living Scale, score of Barthel for Activities of Daily Living score evaluation and SPPB Scale | At inclusion
Evaluation of Cognition with Mini Mental Status Examination (MMSE) | At inclusion
Fragility level (Rockwood criteria) | At inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Marie DANET-LAMASOU, Dr, Principal Investigator — Universitary Hospital
Locations (1):
- University Hospital of Bordeaux - Xavier Arnozan Hospital, Pessac, France